CLINICAL TRIAL: NCT00780780
Title: A Randomized Parallel, Masked to Evaluate the Efficacy of Triamcinolone Associated With Nepafenac (Nevanac) Compared With Intravitreal Injection of Triamcinolone for Treatment of Clinically Significant Diabetic Macular Edema
Brief Title: Efficacy Study of Triamcinolone Associated With Nepafenac for Treatment of Diabetic Macular Edema
Acronym: NEVANAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Rubens Belfort Jr. - Full Professor of Ophthalmology, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 0754/07
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2012-08

CONDITIONS: Diabetic Macular Edema
Keywords: triamcinolone; nepafenac; DME; edema macular
MeSH Terms: conditions — Macular Edema | interventions — Triamcinolone; nepafenac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Triamcinolone intravitreal injection + Nepafenac eye drops
  Interventions: Drug: Triamcinolone + Nepafenac
- 2 (Other): Triamcinolone intravitreal injection
  Interventions: Drug: triamcinolone intravitreal injection

INTERVENTIONS:
Drug: Triamcinolone + Nepafenac — Triamcinolone intravitreal injection 0,1 ml (4mg) Nepafenac 1 drop, tid, during 6 months
  Other Names: Nepafenac (Nevanac)
  Arms: 1
Drug: triamcinolone intravitreal injection — triamcinolone intravitreal injection
  Other Names: triamcinolone
  Arms: 2

SUMMARY:
Diabetics retinopathy remains the major threat to sight in the working age population in the developed world. Furthermore, it is increasing as a major cause of blindness in other parts of the world, especially developing countries. Diabetic macular edema (DME) is a manifestation of diabetic retinopathy that produces loss of central vision.

The triamcinolone intravitreal injection (1-4mg) is indicated to treatment of diabetic macular edema and it is considered an important treatment since it improves the visual acuity of patients with resolution of edema.

Nepafenac is a non-steroidal anti-inflammatory drug (NSAID), usually sold as a prescription eye drop (0.1% solution). Nepafenac is manufactured by Alcon as Nevanac. It is approved by FDA as well as ANVISA. Pre-clinical studies suggest this medication showed efficacy to treat ocular posterior segment inflammation.

The purpose of this study is evaluate the efficacy of intravitreal triamcinolone associated with nepafenac eye drops as treatment of diabetic macular edema.

DETAILED DESCRIPTION:
We plan to enroll 40 patients in this prospective randomized clinical trial. Eligible patients will be randomized into two groups. All patients will have Early Treatment of Diabetic Retinopathy Study (ETDRS) vision measured and OCT (OCT Stratus - Zeiss)in both eyes in following visits: Baseline, Week 4, 8, 12, 20 and 25. OCT measurements will include total macular volume, central foveal thickness, and average macular thickness. The patients will be evaluated during 25 weeks (7 visits). Parameters for clinical evaluation: visual acuity, IOP, biomicroscopy, fundus examination through dilated pupil and OCT.

Group A: 20 patients will receive intravitreal triamcinolone injection Group B: 20 patients will receive intravitreal triamcinolone injection associated with nepafenac eye drops (1 gtt, tid) during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at least
* Diagnosis of diabetes mellitus (type 1 or type 2. any one of the following will be considered to be sufficient evidence that diabetes is present:

  * current regular use of insulin for the treatment of diabetes
  * current regular use of oral hypoglycemic agents for the treatment of diabetes diabetes as defined by american Diabetes Association (ADA)
  * symptoms of diabetes (polyuria, polydipsia, and unexplained weight loss) or eigth-hour fasting plasma glucose > 126 mg/dl
* Diabetic macular edema clinically observable associated with diabetic retinopathy:

  * prior treated with any treatment or one or three sessions focal laser or grid for DME, intervals between sessions must be at least 30 days
  * the most recent laser at least 3 months prior to Baseline, or no prior medical therapy for diabetic macular edema, or in the investigator opinion the patient would not benefit from macular laser treatment, or the patient refuses laser treatments
* BCVA score between 34 letters (20/320 ETDRS)e 68 letters (20/40 ETDRS) in the study eye measured by the ETDRS method at qualification/baseline visit
* Retinal thickness > 250 um by OCT

Exclusion Criteria:

* Uncontrolled systemic disease
* Initiation of medical therapy for diabetes or a change from oral hypoglycemic agents to insulin therapy within 4 months prior to the qualification visit
* Renal failure requiring hemodialysis or peritoneal dialysis within 6 months prior to the qualification visit
* Any ocular condition in the study eye that in the opinion of the investigator would prevent a 15 letters improvement of visual acuity (e.g. severe macular ischemia)
* Presence of branch retinal vein occlusion, central retinal vein occlusion, uveitis, pseudophakic cystoid edema or any other condition in the study eye which could be contributing to macular edema
* Presence of an epiretinal membrane in the study eye
* History of IOP elevation in response to steroid treatment in either eye
* History of glaucoma or optic nerve head change consistent with glaucoma damage, and/or glaucomatous visual field loss in the study eye
* Ocular hypertension in the study eye requiring more than 1 anti-glaucoma medication to maintain IOP < 22mmHg at qualification visit
* Presence of anterior chamber intraocular lens in the study eye
* Active optic disc or retinal neovascularization in the study eye at qualification visit
* Active or history of choroidal neovascularization in the study eye
* Presence of rubeosis irides in the study eye at qualification visit
* Any active ocular infection (i.e. bacterial, viral, parasitic or fungal) in qualification
* History of herpetic infection in the study eye or adnexa
* Presence of active or inactive toxoplasmosis in either eye at qualification
* Presence of visible scleral thinning or ectasia in the study eye
* Media opacity in the study eye at qualification
* Intraocular surgery, including cataract surgery, and/or laser of any type in the study eye within 90 days prior to qualification.
* History of central serous chorioretinopathy in either eye
* History of pars plana vitrectomy in the study eye
* History of use of intravitreal steroids in the study eye within 3 months prior qualification
* Periocular depot of steroids to the study eye with 3 months prior to qualification
* Use of systemic steroids within 1 month prior qualification or anticipated use at any time during the study
* Use of inhibitors of carbonic anhydrase within 1 month prior qualification or anticipated use at any time during the study
* Use of immunosuppressants, immunomodulators, antimetabolites and/or alkylating agents with 6 months prior to qualification or anticipated use at any time during the study
* BCVA < 34 letters (20/200 snellen equivalent) in the non-study eye using the ETDRS at qualification
* Known allergy of hypersensitivity to the study medication or its components
* Known allergy or contraindication to the use of fluorescein or povidone iodine
* Contraindication to pupil dilation in either eye
* Female patients who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Weeks 1, 4, 8, 12, 20 and 25
Optical coherence tomography (OCT) | Weeks 4, 8, 12, 20 and 25

SECONDARY OUTCOMES:
Biomicroscopy/Fundus examination | Day 1, Weeks: 1, 4, 8, 12, 20 and 25

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort Jr, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo - Dept. of Ophthalmology / Vision Institute, São Paulo, São Paulo, Brazil